CLINICAL TRIAL: NCT05198076
Title: The Long Term Efficacy of High Frequency Repetitive Transcranial Magnetic Stimulation on Postural Stability in Parkinsonian Patients.
Brief Title: 6 Month Follow up Study on the Changes of Postural Stability in Parkinsonian Patients in Response to High Frequency TMS.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Engy Badreldin Saleh Moustafa, PhD, Lecturer of P.T for neuromuscular disorders and its surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003448
Record Dates: First submitted 2022-01-02; First posted 2022-01-20 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Double Blind Randomized Control Trial
Who Masked: Participant, Care Provider
Masking Description: Randomization was done using Sealed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G1 ( Conventional Physical Therapy Program group) (No Intervention): Patients in (G1) will be treated by a designed physiotherapy program consisted of aerobic exercise on treadmill, stretching exercise, Proprioceptive neuromuscular facilitation (PNF) techniques, Graduated active exercises, gait training, Reciprocal and weight shifting exercises. The treatment will be conducted three sessions per week, day after day for successive four weeks. The session duration was 40min to 1 hour.
- G2 ( High Frequency rTMS group) (Experimental): Patients in (G2) will be treated by high frequency repetitive transcranial magnetic stimulation (HF-rTMS) in addition to the same physiotherapy program as in G1. The treatment will be conducted three sessions per week, day after day for successive four weeks. The session duration for rTMS will be 20-30 minutes, the physiotherapy session will be 40-45 min.
  Interventions: Device: High Frequency Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: High Frequency Repetitive Transcranial Magnetic Stimulation — The High Frequency repetitive TMS will be delivered to the scalp over the primary motor cortex contralateral to the more affected side using a MAGSTIM rapid2 machine (Model P/N 3576-23-09, MAGSTIM Company LTD, UK) connected with a figure - of- eight shaped coil. Each patient will receive 12 sessions over four weeks. Position of the coil will be adjusted to find the optimal scalp position and the location of stimulation that will be marked to maintain consistency among sessions. The session will consist of 24 trains of 50 stimuli each delivered at five Hz. The procedure will be conducted with the patients in the ''On'' state (75 min. after medications)
  Other Names: HF-rTMS
  Arms: G2 ( High Frequency rTMS group)

SUMMARY:
Postural instability is one of the cardinal signs in Parkinson's disease (PD). It represents one of the most disabling symptoms in the advanced stages of the disease. It is associated with frequent falls and loss of independence. The aim of the current study is to assess the long term efficacy of high frequency repetitive transcranial magnetic stimulation (rTMS) on improving postural instability in PD patients.

DETAILED DESCRIPTION:
Thirty to forty PD patients will be recruited who fulfill the U.K Parkinson's Disease Brain Bank Criteria for idiopathic PD. Patients with mild to moderate disease severity according to UPRS and Modified Hoehn and Yahr staging, age ranged from 55-70 years, duration of illness from two to five years will be included. The patients who will match our inclusion criteria will be assigned randomly into two equal groups; control group (G1) will receive a designed physical therapy program and study group (G2) will receive 12 sessions of (5Hz) rTMS over the primary motor cortex in addition to the same physical therapy program as in G1. The treatment will be conducted three times per week, over four weeks.

Biodex balance system will be used to assess objectively balance indices (overall, anterio-posterior and medio-lateral balance index) and dynamic limit of stability (overall LOS score, time to complete test) pretreatment , posttreatment and one month later as a follow up.

ELIGIBILITY:
Inclusion Criteria:

* All included patients should fulfill the U.K Parkinson's Disease Brain Bank Criteria for idiopathic PD.
* Patients with mild to moderate disease severity according to UPRS and Modified Hoehn and Yahr staging
* Duration of illness from two to five years were included.
* All included patients should be medically and psychologically stable and of adequate cardiac function.
* All included patients should haven't receive any rTMS sessions before.
* Signed consent form should be taken from all included patients.

Exclusion Criteria:

* Patients with implanted devices, serious medical illness or history of seizures were excluded.
* Patients with severe freezing phenomenon or severe tremors were excluded

Ages: 55 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2025-12-18 (Estimated); Study Completion 2026-02-18 (Estimated)

PRIMARY OUTCOMES:
Overall stability index (OSI) | Changes from Pre-intervention to immediately post intervention, Changes from immediately post intervention to six month follow up.
  Biodex Balance System SD (Model 945-302, software version 3.12, New York). The system consists of a circular platform supported. It can tilt 20° in all directions from the horizontal. The system's microprocessor-based actuator controls the extent of the surface instability of the platform. The system will evaluate two components of balance (balance indices and dynamic limit of stability). To assess balance indices; each patient was asked to maintain the center of mass in the middle of a concentric circle that appeared on the screen placed in front of the patient. The instrument records the actual postural sway and calculates the variance from the center, which is expressed as a balance index.
Antero-posterior Stability index (APSI) | Changes from Pre-intervention to immediately post intervention, Changes from immediately post intervention to six month follow up.
  Biodex Balance System SD (Model 945-302, software version 3.12, New York). The system consists of a circular platform supported. It can tilt 20° in all directions from the horizontal. The system's microprocessor-based actuator controls the extent of the surface instability of the platform. The system will evaluate two components of balance (balance indices and dynamic limit of stability). To assess balance indices; each patient was asked to maintain the center of mass in the middle of a concentric circle that appeared on the screen placed in front of the patient. The instrument records the actual postural sway and calculates the variance from the center, which is expressed as a balance index.
Medio-lateral stability index (MLSI) | Changes from Pre-intervention to immediately post intervention, Changes from immediately post intervention to six month follow up.
  Biodex Balance System SD (Model 945-302, software version 3.12, New York). The system consists of a circular platform supported. It can tilt 20° in all directions from the horizontal. The system's microprocessor-based actuator controls the extent of the surface instability of the platform. The system will evaluate two components of balance (balance indices and dynamic limit of stability). To assess balance indices; each patient was asked to maintain the center of mass in the middle of a concentric circle that appeared on the screen placed in front of the patient. The instrument records the actual postural sway and calculates the variance from the center, which is expressed as a balance index.
Directional control percent | Changes from Pre-intervention to immediately post intervention, Changes from immediately post intervention to six month follow up.
  To assess dynamic limit of stability; each patient will be asked to move the center of mass, without changing foot position, into 8 targets (in forward, backward, right ,left, forward-right, forward-left, backward-right, and backward-left direction), the perimeter of which corresponded to 50 percent of the theoretical LOS. The target is displayed on the screen by a blinking square, which appeared randomly in different directions only once. The instrument will calculate the shortest vertical or horizontal path to reach the target from the center in each direction which will be expressed as the directional control score.
Time to complete test | Changes from Pre-intervention to immediately post intervention, Changes from immediately post intervention to six month follow up.
  Each patient will be asked to move the center of mass, without changing foot position, into 8 targets (in forward, backward, right ,left, forward-right, forward-left, backward-right, and backward-left direction), Then the instrument will calculate the time taken to complete each test, the maximum time allowed to perform the movements to complete the LOS test was 300 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Engy BadrEldin S Moustafa, PhD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Ad Doqi, Giza District, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim SD, Allen NE, Canning CG, Fung VS. Postural instability in patients with Parkinson's disease. Epidemiology, pathophysiology and management. CNS Drugs. 2013 Feb;27(2):97-112. doi: 10.1007/s40263-012-0012-3. PMID 23076544
- [Background] Benninger DH, Iseki K, Kranick S, Luckenbaugh DA, Houdayer E, Hallett M. Controlled study of 50-Hz repetitive transcranial magnetic stimulation for the treatment of Parkinson disease. Neurorehabil Neural Repair. 2012 Nov-Dec;26(9):1096-105. doi: 10.1177/1545968312445636. Epub 2012 May 15. PMID 22593114
- [Background] Maruo T, Hosomi K, Shimokawa T, Kishima H, Oshino S, Morris S, Kageyama Y, Yokoe M, Yoshimine T, Saitoh Y. High-frequency repetitive transcranial magnetic stimulation over the primary foot motor area in Parkinson's disease. Brain Stimul. 2013 Nov;6(6):884-91. doi: 10.1016/j.brs.2013.05.002. Epub 2013 May 29. PMID 23769414
- [Background] Brandmeir NJ, Brandmeir CL, Kuzma K, McInerney J. A Prospective Evaluation of an Outpatient Assessment of Postural Instability to Predict Risk of Falls in Patients with Parkinson's Disease Presenting for Deep Brain Stimulation. Mov Disord Clin Pract. 2015 Nov 27;3(2):151-155. doi: 10.1002/mdc3.12257. eCollection 2016 Mar-Apr. PMID 30713907
- [Background] Yang YR, Tseng CY, Chiou SY, Liao KK, Cheng SJ, Lai KL, Wang RY. Combination of rTMS and treadmill training modulates corticomotor inhibition and improves walking in Parkinson disease: a randomized trial. Neurorehabil Neural Repair. 2013 Jan;27(1):79-86. doi: 10.1177/1545968312451915. Epub 2012 Jul 10. PMID 22785003
- [Background] Ganesan M, Sathyaprabha TN, Gupta A, Pal PK. Effect of partial weight-supported treadmill gait training on balance in patients with Parkinson disease. PM R. 2014 Jan;6(1):22-33. doi: 10.1016/j.pmrj.2013.08.604. Epub 2013 Sep 8. PMID 24021298
- [Background] Vadala M, Vallelunga A, Palmieri L, Palmieri B, Morales-Medina JC, Iannitti T. Mechanisms and therapeutic applications of electromagnetic therapy in Parkinson's disease. Behav Brain Funct. 2015 Sep 7;11:26. doi: 10.1186/s12993-015-0070-z. PMID 26347217